CLINICAL TRIAL: NCT02233725
Title: Pilot-Study - Incorporating Contrast-Enhanced Ultrasound (CEUS) to Real-Tim MRI / Ultrasound Fusion Imaging for Prostate Biopsies
Brief Title: MRI / Ultrasound Fusion With Contrast-Enhanced Ultrasound Guidance
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H14-00830
Record Dates: First submitted 2014-08-28; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Neoplasms
Keywords: Prostatic Neoplasms; Magnetic Resonance Imaging; MRI / Ultrasound Fusion; Contrast-Enhanced Ultrasound (CEUS)
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Definity Perflutren Suspension (Active Comparator): Injection of Definity Perflutren Injectable Suspension- which travels in the bloodstream throughout the body. These microbubbles are identifiable on ultrasound imaging, and studies of the liver and kidney have identified it as a useful adjunct to identifying vascular lesions. Areas of regular blood flow will not have as large a concentration of the microbubble agent as will areas that have increased blood flow and neovascularisation. It has been well documented that cancerous solid lesions undergo neovascularisation and have increased blood flow to the area.
  Interventions: Device: Definity Perflutren Injectable Suspension

INTERVENTIONS:
Device: Definity Perflutren Injectable Suspension — a single dose of 10 μL/kg of the activated product by intravenous bolus injection over 30-60 seconds, followed by a 10 mL saline flush. If necessary, a second 10 μL/kg dose may be administered 5 minutes after the first injection to prolong contrast enhancement
  Other Names: Lantheus DEFINITY; FDA Application No. - (NDA) 021064; Active Ingredient(s) - PERFLUTREN; Strength- 6.52MG/ML; Dosage Form/Route - INJECTABLE;INTRAVENOUS

SUMMARY:
Prostate cancer is the most common cancer in men. It is most often detected by an abnormal digital rectal exam or an elevated Prostate-Specific Antigen -determine by a blood test. When it is suspected that someone may have prostate cancer, a biopsy is ordered. This biopsy is performed by the Radiologist with ultrasound guidance through the rectum. In some patients, a Magnetic Resonance Imaging (MRI) scan of the prostate may be ordered to further evaluate the prostate. In some situations, the MRI and Ultrasound images will be fused (digitally merged) together during the ultrasound procedure to help localize the questionable lesions. Recent research has used an additional component known as a contrast agent - an intravenously injected inert substance - which is identifiable by ultrasound. This inert substance is more obvious in areas of increased blood flow, which is a common finding in cancerous lesions. In this research project, we would like to determine whether the use of contrast-enhanced ultrasound is beneficial in improving accuracy of the biopsies taken and the relative correlation to the MRI/ Ultrasound-fused images.

DETAILED DESCRIPTION:
It is the hypothesis that cancerous lesions in the prostate will have an increased amount of blood flow, and that the lesions identified under ultrasound with the benefits of contrast-enhanced imaging can be correlated to the MRI Findings in real-time. A study of 50 patients who would be undergoing MRI/Ultrasound fusion would be selected to have contrast added to their procedure. The lesions identified on MRI would then be evaluated with contrast-enhanced ultrasound. The findings from the contrast study could then be correlated with the MRI findings. The rest of the prostate gland would also be assessed using the contrast agent for lesions not identified on the MRI imaging study. The pathology results could be correlated with both the contrast study and the MRI study both independently, and in conjunction with the two imaging modalities. If a correlation between highly suspicious lesions on the MRI and significant flow patterns under contrast can be established, then the sensitivity and specificity of contrast-enhanced ultrasound can be increased.

While MRI / Ultrasound Fusion is being shown to increase prostate cancer identification and targeting for biopsy, it is a very limited modality due to the costs associated. Many sites will also not have access to an MRI unit, and the fusion system is prohibitively expensive, and requires specialized training to configure the system and modulate the images in real-time. However, ultrasound is an in expensive modality that is readily available. If the materials and methods in the utilization of contrast-enhanced ultrasounds can be correlated to MRI / Ultrasound fusion, better protocols can be developed for contrast-enhanced ultrasound. This more cost-effective method of identifying and targeting prostate cancer could then be exported to smaller communities who would otherwise still be carrying out the sextant biopsy model.

ELIGIBILITY:
Inclusion Criteria:

* Adults ( aged 21 years or greater), English speaking patients

Exclusion Criteria:

* Patients who are unable to provide informed consent
* Patients who have had previous reaction to any contrast agent at any point in the past
* Patients who have had previous septic infection from prostate biopsies at any point in the past
* Patients who have a right-to-left, bi-directional, or transient right-to-left cardiac shunts.
* Patients undergoing extracorporeal shock wave lithotripsy for urinary calculi.
* Patients with pre-existing cardiopulmonary compromise including, but not limited to, acute myocardial infarction, acute coronary artery syndromes, worsening or unstable congestive heart failure, serious ventricular arrhythmias or respiratory failure, including patients receiving mechanical ventilation

Min Age: 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Measure the quality and pathology results of prostate samples taken during Contrast-Enhanced Ultrasound (CEUS) with MRI/ Ultrasound fusion. | 1 Day
  It is hypothesized that the introduction of the Definity contrast agent during the ultrasound biopsy will increase the accuracy of the targeting biopsy sample, as well as reduce the number of targeted biopsies of non-cancerous lesions. We will compare the MRI characteristics of the prostate lesions in question in real-time ( as the MRI and Ultrasound will be fused together ), and determine whether questionable lesions seen under MRI have increased flow dynamics

SECONDARY OUTCOMES:
Measure whether the use of Contrast-Enhanced Ultrasound (CEUS) on prostate cancer detection rates when incorporated with MRI / Ultrasound Fusion differs from non-CEUS prostate biopsies performed under MRI/ Ultrasound Fusion guidance | 1 Day
  We will measure the number of prostate samples that are determined to be positive for prostate cancer, and compare that with a control group with similar prostate characteristic appearances.

OTHER OUTCOMES:
Generate a Time Intensity Curve for prostate cancer lesions and measure the relation of that value to the MRI Apparent Diffusion Coefficient (ADC) value of the lesion. | 1 month
  Ultrasound Contrast enhancement has a time component, and the measuring of the contrast uptake as a function of time will be measured to generate a Time Intensity Curve (TIC). The time to the contrast enhancement peak (TTP), intensity change from the baseline to peak (ΔI) and ΔI/TTP of the tumour and the the TIC will be correlated to the lesion's MRI Apparent Diffusion Coefficient (ADC) value.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Eddy, BSc, Study Director — VCH
Locations (1):
- Vancouver Coastal Health (VCHRI/VCHA), Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Maxeiner A, Fischer T, Stephan C, Cash H, Slowinski T, Kilic E, Durmus T. [Real-time MRI/US fusion-guided biopsy improves detection rates of prostate cancer in pre-biopsied patients]. Aktuelle Urol. 2014 May;45(3):197-203. doi: 10.1055/s-0034-1375682. Epub 2014 Jun 5. German. PMID 24902069
- [Background] Rifkin MD, Dahnert W, Kurtz AB. State of the art: endorectal sonography of the prostate gland. AJR Am J Roentgenol. 1990 Apr;154(4):691-700. doi: 10.2214/ajr.154.4.1690499. No abstract available.
- [Background] Oyen R, Van Popel H, Van de Voorde W, Knapen P, Ameye F, Baert AL, Baert LV. [The significance of focal hypoechoic lesions in the peripheral zone of the prostate]. J Belge Radiol. 1995 Dec;78(6):356-8. Dutch. PMID 8576025
- [Background] Sibley RI, Sibley AF. Correlation of digital rectal examination, prostate specific antigen, and transrectal ultrasound in prostate carcinoma in African Americans. J Natl Med Assoc. 1997 May;89(5):318-23. PMID 9170832
- [Background] Norberg M, Egevad L, Holmberg L, Sparen P, Norlen BJ, Busch C. The sextant protocol for ultrasound-guided core biopsies of the prostate underestimates the presence of cancer. Urology. 1997 Oct;50(4):562-6. doi: 10.1016/S0090-4295(97)00306-3. PMID 9338732
- [Background] Halpern EJ, Ramey JR, Strup SE, Frauscher F, McCue P, Gomella LG. Detection of prostate carcinoma with contrast-enhanced sonography using intermittent harmonic imaging. Cancer. 2005 Dec 1;104(11):2373-83. doi: 10.1002/cncr.21440. PMID 16240450
- [Background] Mitterberger M, Pinggera GM, Horninger W, Bartsch G, Strasser H, Schafer G, Brunner A, Halpern EJ, Gradl J, Pallwein L, Frauscher F. Comparison of contrast enhanced color Doppler targeted biopsy to conventional systematic biopsy: impact on Gleason score. J Urol. 2007 Aug;178(2):464-8; discussion 468. doi: 10.1016/j.juro.2007.03.107. Epub 2007 Jun 11. PMID 17561137